CLINICAL TRIAL: NCT04579159
Title: Multicentre, Intern., Inv.-Initiated, Single-arm Case-finding Study of a Cloud Based Analytic Service as Screening Tool to Detect and Quantify Episodes of Absolute Arrhythmia Using an Automated, Wearable PPG-based Monitoring System
Brief Title: The Smartphone and Wearable Detected Atrial Arrhythmia in Older Adults Case Finding Study (Smart in OAC - AFNET 9)
Acronym: Smart in OAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atrial Fibrillation Network (Other)
Collaborators: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry); Preventicus GmbH (Industry); Corsano/ MMT (Unknown); Getemed Medizin- und Informationstechnik (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Smart in OAC - AFNET 9
Record Dates: First submitted 2020-09-08; First posted 2020-10-08 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Atrial Arrhythmia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- only control group (Other): To investigate the specificity of the wearable and to gather more information on ECG abnormalities in the population studied, a randomly selected group of participants without wearable-detected AA within 8 weeks of screening (same number as screen-positives and verified by Telecare) will also be invited to obtain a 14day Tele ECG (patch).
  Interventions: Device: Preventicus heartbeat app in combination with wearables

INTERVENTIONS:
Device: Preventicus heartbeat app in combination with wearables — CE certified devices

SUMMARY:
This feasibility study will develop and evaluate pathways to identify participants with wearable-detected absoulute Arrhythmia (AA) and to enable local study teams to contact them regarding participation in a controlled trial of oral anticoagulation in this population, which will be conducted after the feasibility study.

DETAILED DESCRIPTION:
In this study, the feasibility of evaluating the efficacy of a cloud based analytic service in combination with a PPG-wearable in detecting AA will be assessed and the number of cases found. The design aims to provide simple, low-threshold access to this screening technology targeting at-risk populations. This study will not cause any restrictions on the usual care of the study participants. Access to the screening will be provided close to home and free of charge. The app will also be used to validate and enhance the clinical information about the participants captured during the study. This information will be used to define and refine target groups with highest screening efficiency and, in the long-term, outcome benefits. The study will describe the prevalence of AA in an unselected population that can be reached by a low-threshold screening procedure. The study will also generate important information on the different possible screening environments in different countries (e.g. pharmacies, GP practices, etc). Structures of work-up and continuous patient management in screen-positive individuals will be described and may help to design screening pathways in the main trial. By verifying the wearable-diagnoses by ECG in all screen-positive and a random selection of screen-negative participants, the diagnostic accuracy of the wearable in combination of cloud based analytic service can be estimated. Cost effectiveness assessment will evaluate the cost of low-threshold remote screening per patient identified and help guide to target high risk groups with optimal screening yield in the future. The collected data will provide the sound basis for the design and conduct of a large outcome trial.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* 65 years or older
* Willing and able to provide informed consent
* Owning mobile phone compatible with the PPG-wearable

Exclusion criteria:

* Known AF
* Known current or planned oral anticoagulation treatment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 882 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with newly detected AA within 4 weeks of device use of all participants included in the study | Screening per participant: 4-8 weeks
  Proportion of participants with newly detected AA within 4 weeks of device use of all participants included in the study

SECONDARY OUTCOMES:
Propotion of participants with AA detected at any time, including those with AA detected within the full time of recording | Screening per participant: 4-8 weeks ECG screening: 2 weeks Overall study duration: 12 months
  Propotion of participants with AA detected at any time, including those with AA detected within the full time of recording
Time from completed enrolment to the first positive screening, taking death as compeeting risk into account | Screening per participant: 4-8 weeks ECG screening: 2 weeks Overall study duration: 12 months
  Time from completed enrolment to the first positive screening, taking death as compeeting risk into account
Regional differences of AA prevalance (diagnostic yield) | Screening per participant: 4-8 weeks ECG screening: 2 weeks Overall study duration: 12 months
  Regional differences of AA prevalance (diagnostic yield)
Differences by rout fo invitation and enrolment | Screening per participant: 4-8 weeks ECG screening: 2 weeks Overall study duration: 12 months
  Differences by rout fo invitation and enrolment
Duration of atrial arrhythmia episodes | Screening per participant: 4-8 weeks ECG screening: 2 weeks Overall study duration: 12 months
  Duration of atrial arrhythmia episodes will be reported descriptively by mean, sd, range, median and IQR
Follow-up EQ-5DL-5L viscual analogue scale of participants with positve PPG | Screening per participant: 4-8 weeks ECG screening: 2 weeks Overall study duration: 12 months
  Follow-up EQ-5DL-5L viscual analogue scale of participants with positve PPG
Detection of AF: Number of participants with clinically confirmed arrhythmias during Holter ECG | Screening per participant: 4-8 weeks ECG screening: 2 weeks Overall study duration: 12 months
  Detection of AF: Number of participants with clinically confirmed arrhythmias during Holter ECG, documented clinically or by event-recorder
Compliance: The compliance of participants with protocol with regards to the measurement procedure of the app and wearable | Screening per participant: 4-8 weeks ECG screening: 2 weeks Overall study duration: 12 months
  Compliance: The compliance of participants with protocol with regards to the measurement procedure of the app and wearable will be presented descriptively

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Fabritz, Professor, Principal Investigator — Institute of Cardiovascular Sciences, University of Birmingham
Locations (4):
- Germany (2):
  - Universitäres Herz- und Gefäßzentrum UKE Hamburg, Hamburg
  - Kardiologische Praxis, Dr. med. Jens Taggeselle, Markkleeberg
- Krakowskie Centrum Diagnostyczno-Kliniczne (KCDK), Krakow, Poland
- Hospital Clínic Unitat d'Arrítmies, Institut Cardiovascular, Barcelona, Catalonia, Spain

REFERENCES:
- [Derived] Fabritz L, Connolly DL, Czarnecki E, Dudek D, Guasch E, Haase D, Huebner T, Zlahoda-Huzior A, Jolly K, Kirchhof P, Obergassel J, Schotten U, Vettorazzi E, Winkelmann SJ, Zapf A, Schnabel RB; Smart in OAC-AFNET 9 investigators. Smartphone and wearable detected atrial arrhythmias in Older Adults: Results of a fully digital European Case finding study. Eur Heart J Digit Health. 2022 Nov 1;3(4):610-625. doi: 10.1093/ehjdh/ztac067. eCollection 2022 Dec. PMID 36710894
- [Derived] Fabritz L, Connolly D, Czarnecki E, Dudek D, Zlahoda-Huzior A, Guasch E, Haase D, Huebner T, Jolly K, Kirchhof P, Schotten U, Zapf A, Schnabel RB. Remote Design of a Smartphone and Wearable Detected Atrial Arrhythmia in Older Adults Case Finding Study: Smart in OAC - AFNET 9. Front Cardiovasc Med. 2022 Mar 21;9:839202. doi: 10.3389/fcvm.2022.839202. eCollection 2022. PMID 35387433